CLINICAL TRIAL: NCT06335134
Title: A Single-Center, Open-Label Study to Evaluate the Effect of XW003 Injection on the Pharmacokinetics of Metformin, Warfarin, Rosuvastatin or Digoxin in Healthy Subjects
Brief Title: A Drug-Drug Interaction Study Between XW003 and Metformin, Warfarin, Rosuvastatin or Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SCW0502-1016
Record Dates: First submitted 2023-07-29; First posted 2024-03-28 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers
Keywords: Ecnoglutide; XW003; Metformin; Warfarin; Rosuvastatin; Digoxin
MeSH Terms: interventions — Metformin; Warfarin; Rosuvastatin Calcium; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trial Group 1: Metformin and Warfarin administered before and with XW003 treatment (Experimental): Metformin will be dosed twice daily (0.5 mg per dose) in two periods of 3.5 days for a total of 7 doses before and with XW003 treatment. Single doses of warfarin (2.5 mg per dose) will be given before and with XW003 treatment. The two drugs will be separated by a washout. XW003 will be administered subcutaneously once weekly in escalating doses of 0.3 mg for 4 weeks, 0.6 mg for 4 weeks and 1.2 mg for 4 weeks.
  Interventions: Drug: XW003 injection; Drug: Metformin; Drug: Warfarin
- Trial Group 2: Rosuvastatin and Digoxin administered before and with XW003 treatment (Experimental): Single doses of rosuvastatin (10 mg per dose) and digoxin (0.25 mg per dose) will be given before and with XW003 treatment. The two drugs will be separated by a washout. XW003 will be administered subcutaneously once weekly in escalating doses of 0.3 mg for 4 weeks, 0.6 mg for 4 weeks and 1.2 mg for 4 weeks.
  Interventions: Drug: XW003 injection; Drug: Rosuvastatin; Drug: Digoxin

INTERVENTIONS:
Drug: XW003 injection — Administered subcutaneously
  Other Names: ecnoglutide
Drug: Metformin — Administered orally
  Arms: Trial Group 1: Metformin and Warfarin administered before and with XW003 treatment
Drug: Warfarin — Administered orally
  Arms: Trial Group 1: Metformin and Warfarin administered before and with XW003 treatment
Drug: Rosuvastatin — Administered orally
  Arms: Trial Group 2: Rosuvastatin and Digoxin administered before and with XW003 treatment
Drug: Digoxin — Administered orally
  Arms: Trial Group 2: Rosuvastatin and Digoxin administered before and with XW003 treatment

SUMMARY:
This is a study of a drug-drug interaction between XW003 and Metformin, Warfarin, Rosuvastatin or Digoxin

DETAILED DESCRIPTION:
This is a single-center, open-label, fixed-sequence study designed to assess the effect of once-weekly subcutaneous injections of XW003 on the pharmacokinetics of metformin, warfarin, rosuvastatin or digoxin. Approximately 56 healthy subjects are to be enrolled into 2 parallel trial groups, with 28 subjects and 2 drugs evaluated in each of the trial group

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-45 years old, inclusive;
2. BMI: 20.0 to 30.0 kg/m2 , body weight: ≥50.0kg.
3. Ability and willingness to participate in the study, give written informed consent, and comply with the study requirements and all protocol procedures.

Exclusion Criteria:

1. Presence of clinically significant conditions (including but not limited to respiratory system, cardiovascular system, gastrointestinal system, endocrine system, immune system, integumentary system, nervous system, ENT or other related diseases);
2. History of allergic diseases including asthma, urticaria or eczema, or history of sensitivity to GLP-1 products, digoxin, warfarin, rosuvastatin or metformin;
3. Known difficulty in swallowing tablets or history of gastrointestinal diseases affecting drug absorption;
4. History of receiving any procedures that might affect drug absorption, distribution, metabolism or excretion;
5. History of acute or chronic pancreatitis;
6. History of documented or suspected hypoglycemic episodes within 6 months prior to screening;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of metformin: AUC0-inf | up to 101 days
Pharmacokinetics of S-warfarin and R-warfarin: AUC0-inf | up to 114 days
Pharmacokinetics of rosuvastatin: AUC0-inf | up to 102 days
Pharmacokinetics of digoxin: AUC0-inf | up to 112days

CONTACTS AND LOCATIONS:
Overall Officials: Qin Yu, Principal Investigator — West China Second University Hospital
Locations (1):
- West China Second University Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No